CLINICAL TRIAL: NCT04769453
Title: Multicenter Ab-interno Glaucoma Study Investigating Canaloplasty, Randomized, Controlled Trial: iTrack (Nova Eye Medical) Compared to Omni (Sight Sciences)
Brief Title: Multicenter Ab-interno Glaucoma Study Investigating Canaloplasty
Acronym: MAGIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor-initiated, suspension of study due to modification of key parameters.
Sponsor: Nova Eye, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NE 01021
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Canaloplasty
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- iTrack canaloplasty microcatheter with Healon GV Pro (Active Comparator): Patients will be randomized to the iTrack microcatheter (canaloplasty) with Healon GV Pro (ophthalmic viscoelastic device)
  Interventions: Device: Canaloplasty using the iTrack microcatheter with Healon GV Pro
- OMNI surgical system with Healon GV Pro (Active Comparator): Patients will be randomized to the OMNI surgical system (canaloplasty) with Healon GV Pro (ophthalmic viscoelastic device)
  Interventions: Device: Canaloplasty using the Omni surgical system with Healon GV Pro
- iTrack canaloplasty microcatheter with Healon Pro (Active Comparator): Patients will be randomized to the iTrack microcatheter (canaloplasty) with Healon Pro (ophthalmic viscoelastic device)
  Interventions: Device: Canaloplasty using the iTrack microcatheter with Healon Pro
- OMNI surgical system with Healon Pro (Active Comparator): Patients will be randomized to the OMNI surgical system (canaloplasty) with Healon Pro (ophthalmic viscoelastic device)
  Interventions: Device: Canaloplasty using the Omni surgical system with Healon Pro

INTERVENTIONS:
Device: Canaloplasty using the iTrack microcatheter with Healon GV Pro — 360 degree microcatheterization and viscodilation of Schlemm's canal
  Arms: iTrack canaloplasty microcatheter with Healon GV Pro
Device: Canaloplasty using the Omni surgical system with Healon GV Pro — 360 degree microcatheterization and viscodilation of Schlemm's canal
  Arms: OMNI surgical system with Healon GV Pro
Device: Canaloplasty using the iTrack microcatheter with Healon Pro — 360 degree microcatheterization and viscodilation of Schlemm's canal
  Arms: iTrack canaloplasty microcatheter with Healon Pro
Device: Canaloplasty using the Omni surgical system with Healon Pro — 360 degree microcatheterization and viscodilation of Schlemm's canal
  Arms: OMNI surgical system with Healon Pro

SUMMARY:
A prospective, multicenter, randomized, single-masked clinical trial to evaluate the effectiveness outcomes of canaloplasty performed as a standalone procedure with the iTrack microcatheter to the Omni surgical system, and to compare the effectiveness of two types of Ophthalmic Viscoelastic Device (OVD).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with mild to moderate open angle Glaucoma.
2. Visual Field test (Humphrey SITA standard 24-2) with mean deviation better than or equal to -12.0 dB
3. IOP < or = to 36 mmHG while on one to four ocular hypotensive medications
4. Shaffer grade of > or = III in all four quadrants
5. Able and willing to comply with the Protocol and follow up visits for 12 months

Exclusion Criteria:

1. Laser trabeculoplasty other than selective laser trabeculoplasty (SLT)
2. History of iStent or iStent inject within 180 days of the screening visit
3. History of ECP or Micropulse laser
4. Trabeculectomy or other bleb forming procedure including Xen, Express and glaucoma drainage device/valves
5. Prior canaloplasty (ab interno and ab externo)
6. Prior goniotomy or trabeculotomy
7. History of Hydrus microstent or suprachoroidal stent
8. History of cataract surgery within 6 months of screening
9. Acute angle closure, traumatic, congenital, malignant, uveitic or neovascular glaucoma, pigmentary or pseudoexfoliative glaucoma

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Reduction in mean Intraocular pressure (IOP) and glaucoma medication use at 12 months post-intervention | 12 months
  IOP will be measured at each study visit using Goldmann applanation tonometry

SECONDARY OUTCOMES:
Complications intra-operatively and post-operatively associated with the iTrack canaloplasty microcatheter compared to complications intra-operatively and post-operatively with the OMNI surgical system. | 12 months
Visual acuity at 12 months compared to baseline visual acuity | 12 months
  Best corrected visual acuity (BCVA) will be assessed using the standard Snellen eye chart

CONTACTS AND LOCATIONS:
Overall Officials: Shamil Patel, MD, MBA, Principal Investigator — Eye Physicians and Surgeons of Arizona
Locations (7):
- United States (7):
  - Arizona Advanced Eye Research Institute, Glendale, Arizona
  - Beverly Hills Institute of Ophthalmology, Beverly Hills, California
  - Coastal Vision, Orange, California
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Cataract and Laser Institute of Southern Oregon, Medford, Oregon
  - El Paso Eye Surgeons, El Paso, Texas
  - Eye Centers of Racine and Kenosha, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No